CLINICAL TRIAL: NCT07080359
Title: Isavuconazole in Critically Ill Patients: A Study on Antifungal Efficacy and Safety
Brief Title: Isavuconazole in Critically Ill Patients: Efficacy and Safety
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-Xiang Cao, Senior Clinical Pharmacist, Shanghai 10th People's Hospital
Other Study IDs: SHSY-IEC-6.0/25K114/P01
Record Dates: First submitted 2025-06-25; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Fungal Infection; Aspergillosis; Mucormycosis
MeSH Terms: conditions — Mycoses; Aspergillosis; Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Isavuconazole group: Critically ill patients who meet the indicated conditions per the prescribing information, administer isavuconazole as follows: Loading dose: 200 mg every 8 hours (q8h) for three times, Maintenance dose: 200 mg once daily (qd)
  Interventions: Drug: Isavuconazole treatment

INTERVENTIONS:
Drug: Isavuconazole treatment — Administer isavuconazole as follows: Loading dose: 200 mg every 8 hours (q8h) for three times, Maintenance dose: 200 mg once daily (qd)

SUMMARY:
Due to factors such as disease status, gastrointestinal conditions, commonly used medications (e.g., vasopressors), and cardiac output, the plasma concentration of isavuconazole in critically ill patients may differ from that in healthy individuals, exhibiting significant variability.

This study aims to explore the variability of isavuconazole plasma concentrations in critically ill patients and its correlation with efficacy and adverse effects. The research includes:

1. The distribution and variability of isavuconazole plasma concentrations in critically ill patients;
2. Clinical outcomes;
3. Adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult critically ill patients (≥18 years) admitted to ICU with suspected or confirmed invasive fungal infection (IFI)
* IFI diagnosis per EORTC/MSGERC 2019 criteria

Exclusion Criteria:

* Drug allergy
* Inherited short QT syndrome
* Contraindications for nasogastric/oral drug delivery
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients meeting criteria for isavuconazole therapy according to the '2023 Isavuconazole Clinical Expert Consensus'
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiological Progress in Pulmonary Fungal Infections | At treatment day 42
  A chest CT uses X-ray tomography, where the patient lies on a table while the machine rotates to capture cross-sectional images
Plasma concentration | On or after day 7 post-dose
  Venous blood samples were collected, centrifuged to obtain supernatant, and concentrations were measured by liquid chromatography-tandem mass spectrometry
Change in immune function profiles (cellular and humoral immunity markers) | Enrollment (Baseline) → Treatment Day 42
  Specific immune markers (e.g., CD4+/CD8+ counts, immunoglobulin levels, or cytokine profiles) will be selected based on emerging evidence or preliminary data prior to finalizing the statistical analysis plan.
Composite infection biomarker profile (including PCT, CRP, IL-6 and WBC) | Enrollment (Baseline) → Treatment Day 42
  The assessment of infection progression is conducted through a comprehensive scoring system as follows:
  Infection Biomarker Score (0-8 points) based on:
  * PCT >0.5 ng/mL (2 point)
  * CRP >10 mg/L (1 point)
  * IL-6 >30 pg/mL (2 point)
  * WBC >10×10⁹/L (3 point)

SECONDARY OUTCOMES:
Electrocardiogram QT Interval | On day 10 post-dose
  A 6-lead ECG was performed.
Composite liver function outcome (including ALT, AST, bilirubin, ALP, and albumin). | From enrollment (Day 0) through Treatment Day 42
  Hepatic function will be assessed using a composite scoring system (0-10 points) incorporating:
  ALT elevation >3×ULN (2 points) AST elevation >3×ULN (2 points) Total bilirubin >2×ULN (3 points)
  * ALP >2×ULN (2 points)
  * Albumin <3.0 g/dL (1 point)

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through Corresponding author's email upon reasonable request to the corresponding author, subject to privacy/ethical restrictions
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Data will be made available through Corresponding author's email upon reasonable request to the corresponding author, subject to privacy/ethical restrictions